CLINICAL TRIAL: NCT01394744
Title: Determination of Metal Ion Levels in the Serum and Assessment of the Respective Cytokine Production of Peripheral Blood Cells in Patients With a Hard-on-hard Bearing Total Hip Replacement
Brief Title: Determination of Metal Ion Serum Levels and Cytokines in Total Hip Replacement
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: ARCUS-Sportklinik (Unknown); DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Peter Thomas, Prof. Dr., Ludwig-Maximilians - University of Munich
Other Study IDs: 10-1739 / IIS2009029
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Hip Replacement Arthroplasty
Keywords: metal; ion; cytokine; hip arthroplasty; blood; Assessment; cytokine profile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum samples for metal ion and cytokine measurement; blood cells for cytokine-RNA assessment
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the study is the analysis of metal ion serum concentrations and of the cytokine production in the blood of patients with a conventional cementless total hip replacement. The rationale is that a) the bearing wear releases particles respectively metal ions into the joint and the blood which will differ in quantity and composition; b) the cytokine production of peripheral blood mononuclear cells (PBMC) might be influenced to a varying degree by the metal and the ceramic particles.

The patients from whom the respective samples will be analyzed are randomized in one of the following three groups: metal-on-metal, ceramic-on-ceramic or ceramic-on-metal. A 36mm bearing is used in all patients. In this separate study, follow-up data of the clinical and radiographic examinations of the patients are available.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years, necessity of hip replacement, informed consent

Exclusion Criteria:

* acute inflammatory disease, renal disease, other cobalt-chromium implant, ager over 75 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: total of 30 subjects; 10 with metal-on-metal, 10 with ceramic-on-ceramic and 10 with ceramic-on-metal hip replacement;
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2018-11 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Thomas, Prof., Principal Investigator — Ludwig-Maximilans-University
Locations (2):
- Germany (2):
  - Ludwig-Maximilians-University Munich, Dept. of Dermatology, Munich, Bavaria
  - ARCUS Sportklinik, Pforzheim